CLINICAL TRIAL: NCT03623841
Title: Effects of Dual-task Training With Exergame and Treadmill on Executive Function, Dual-task Performance and Cortical Activation in Individuals With Parkinson's Disease and Stroke
Brief Title: Training With Exergame and Treadmill on Executive Function and Dual-task Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17MMHIS193
Record Dates: First submitted 2018-07-29; First posted 2018-08-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Parkinson's Disease; Stroke
Keywords: Executive function; Dual-task performance; Dual-task training
MeSH Terms: conditions — Parkinson Disease; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-task training group (Experimental): Participants in dual-task training group will execute dual-task training via exer-game which combined with treadmill, 3 times per week, least 8 weeks.
  Interventions: Other: Dual-task training
- Treadmill training group (Active Comparator): Participants in treadmill training group will do treadmill training only, 3 times per week, least 8 weeks.
  Interventions: Other: Treadmill training

INTERVENTIONS:
Other: Dual-task training — Participants in experimental group will do dual-task training via exer-game which combined with treadmill
  Arms: Dual-task training group
Other: Treadmill training — Participants in control group will do treadmill training only
  Arms: Treadmill training group

SUMMARY:
This study aimed to investigate the effects of dual-task training with exergame and treadmill on executive function and dual-task performance in individuals with PD and stroke and discuss the correlation between the change values of executive function and dual-task performance after training. Besides, investigate cortical activation after training.

DETAILED DESCRIPTION:
Background: In daily living, walking usually combines with cognitive or motor dual tasks. For individuals with Parkinson's disease (PD), gait performance becomes worse while doing dual tasks, which may due to insufficient executive function. Declined executive function may occur in early stage of PD. For those with stroke, impaired dual-task performance also exists. Although 75% of patients with stroke may suffer from impaired executive function, impaired dual-task performance correlates with declined executive function directly or not still unknown. Undoubtedly, impaired executive function decreases their daily activities. Recently, dual-task training by walking with secondary tasks resulted in improvement of single or dual-task gait performance in individuals with PD. As for stroke, dual-task training performed in walking with secondary tasks and resulted in improvement of single or dual-task gait performance. However, previous studies less mentioned about combine cognitive and motor tasks simultaneously with gait training. While dual-task training with exergame and treadmill can include cognitive and motor tasks simultaneously while walking. Thus, whether dual-task training with exergame and treadmill can improve executive function and dual-task performance in individuals with PD and stroke is worth to investigate. Purposes: To investigate the effects of dual-task training with exergame and treadmill on executive function and dual-task performance in individuals with PD and stroke and discuss the correlation between the change values of executive function and dual-task performance after training. Besides, investigate cortical activation after training. Methods: This research will be implemented in two phases. First phase will include 50 subjects with PD and the second phase will include 50 subjects with stroke. After pre-test, subjects will be randomly assigned into either the experimental group or the control group. Subjects in the experimental group will receive 24 sessions dual-task training with exergame and treadmill in 8 weeks; while the control group will receive treadmill training only in same frequency. Each session lasts an hour. Primary outcomes include general cognitive performance, executive function, dual-task performance, dual-task effects and cortical activation. Secondary outcomes include single walking performance, functional walking and quality of life. Statistical analysis: Descriptive statistics will be generated for all variables. Intergroup differences among baseline characteristics will be evaluated by independent t test or χ2 analysis. Primary and secondary outcomes will be analyzed by two-way repeated measures ANOVA and post-hoc test. The correlation between change values of executive function and dual-task performance will be evaluated by Pearson correlation coefficient. Statistical significance will set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as PD and Hoehn and Yahr stage between 1~3
* Age between 50 to 80
* Able to walk 10 m independently without an assistive device
* A score of greater than or equal to 24 on the mini-mental state examination (MMSE)
* In stable medical condition allowing participation in the testing protocol and intervention

Exclusion Criteria:

* Any comorbidity or disability other than PD that would preclude gait training
* Any uncontrolled health condition for which exercise was contraindicated
* Any neurological or orthopedic disease that might interfere with the study
* Server freezing of gait, FOG questionnaire > 15

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Dual-task walking performance | Change from baseline at 8 weeks
  To evaluate gait parameters while doing dual-task walking

SECONDARY OUTCOMES:
Single walking performance | Change from baseline at 8 weeks
  To evaluate gait parameters while doing single walking
Timed up and go test | Change from baseline at 8 weeks
  To evaluate functional walking ability
Parkinson's Disease Questionnaire 39 | Change from baseline at 8 weeks
  To evaluate the quality of life
Frontal lobe battery test-Chinese version | Change from baseline at 8 weeks
  To evaluate executive function
Trail-making test | Change from baseline at 8 weeks
  To evaluate executive function
Stroop color and word test-Chinese version | Change from baseline at 8 weeks
  To evaluate executive function
Verbal fluency test-Chinese version | Change from baseline at 8 weeks
  To evaluate executive function
Digit span test | Change from baseline at 8 weeks
  To evaluate executive function
Dual-task effects/ costs | 2 months
  to compare the cost between doing dual task and single task
Functional near-infrared spectroscopy | Change from baseline at 8 weeks
  To evaluate the changes of blood perfusion in frontal lobe

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming university, Taipei, Taiwan

REFERENCES:
- [Derived] Zhou JH, Wang RY, Liu YT, Cheng SJ, Liu HH, Yang YR. Effects of dual-task training on gait variability in individuals with Parkinson's disease: A randomized controlled trial. J Sci Med Sport. 2025 Dec;28(12):1012-1018. doi: 10.1016/j.jsams.2025.06.009. Epub 2025 Jun 20. PMID 40610273